CLINICAL TRIAL: NCT03268746
Title: Clinical Investigation of the Visual Outcomes and Safety After Bilateral Implantation of a Trifocal Presbyopia Correcting IOL in a Korean Population
Brief Title: Clinical Investigation of the Visual Outcomes and Safety of a Trifocal Intraocular Lens (IOL) in a Korean Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILH297-P004
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Cataract; Presbyopia
Keywords: Korea; Trifocal; PanOptix; Bilateral implantation; Cataract; Prospective; Single Arm; ACRYSOF; Model TFNT00
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Multifocal IOL (Experimental): AcrySof IQ PanOptix Multifocal IOL Model TFNT00 implanted in the capsular bag following cataract removal. Both eyes will be implanted.
  Interventions: Device: AcrySof IQ PanOptix Multifocal IOL

INTERVENTIONS:
Device: AcrySof IQ PanOptix Multifocal IOL — AcrySof IQ PanOptix Multifocal IOL Model TFNT00 for near, intermediate, and distance vision intended for long-term use over the lifetime of the cataract subject
  Other Names: Model TFNT00; AcrySof® IQ PanOptix™

SUMMARY:
The purpose of this study is to confirm the effectiveness of the investigational lens in a Korean population, especially for visual performance, quality of vision, and subject satisfaction with the visual outcome, as well as the safety of the lens. This trial will be conducted in Korea.

DETAILED DESCRIPTION:
Both eyes of a subject must require cataract surgery to qualify for enrollment into this study. Subjects participating in the trial will attend a total of 9 study visits over a 4-5-month period. Of these 9 visits, 1 is preoperative, 2 are operative, and the remaining 6 are postoperative visits. Primary endpoint data will be collected at the Month 3 visit (Day 90-120 post second eye implantation). The second eye implantation will occur 2-30 days after the first implantation.

ELIGIBILITY:
Inclusion Criteria:

* Requires cataract extraction in both eyes
* Clear intraocular media other than cataracts in both eyes
* Calculated lens power between +16.0 and +24.0 diopter (D)
* Preoperative OR expected postoperative regular corneal astigmatism of < 1.00 D.

Exclusion Criteria:

* Pregnant or lactating
* Any clinically significant corneal abnormality, per the Investigator's expert medical opinion
* Previous corneal transplant; previous ocular trauma; previous refractive surgery
* History of, concurrent, or predisposition to retinal conditions, such as diabetic retinopathy, diabetic macular edema, or macular degeneration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (2):
- South Korea (2):
  - Alcon Investigative Site, Seongnam-si
  - Alcon Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TI, Chung TY, Kim MJ, Lee K, Hyon JY. Visual outcomes and safety after bilateral implantation of a trifocal presbyopia correcting intraocular lens in a Korean population: a prospective single-arm study. BMC Ophthalmol. 2020 Jul 15;20(1):288. doi: 10.1186/s12886-020-01549-z. PMID 32669090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study centers located in Korea.
Pre-assignment Details: Of the 52 enrolled, 7 subjects exited as screen failures prior to implantation. This reporting group includes all implanted subjects (45).
Groups:
- TFNT00: AcrySof IQ PanOptix Multifocal intraocular lens (IOL) Model TFNT00 implanted in the capsular bag following cataract removal. Both eyes were implanted
Period: Overall Study
Arm/Group | TFNT00
Started (Attempted Implantation) | 45
Completed | 44
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This analysis population included all subjects with attempted IOL implantation (successful or aborted after contact with the eye) (Safety Analysis Set).
Groups:
- TFNT00: AcrySof IQ PanOptix Multifocal IOL Model TFNT00 implanted in the capsular bag following cataract removal. Both eyes were implanted
Arm/Group | TFNT00
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 45
  Race: Others | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Korean | 45
  Ethnicity: Others | 0

OUTCOME MEASURES:

1. Primary Outcome: Binocular Defocus Curve at Month 3
Description: The defocus curve (an indicator of the expected range of vision with a presbyopia-correcting IOL) was tested binocularly (both eyes together) with the subject's best distance correction across full range varied from +2.0 diopter (D) to -5.0 D in 0.5 D increments. The visual acuity (VA) at each spherical power was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A lower numeric value represents better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 (Day 90-120 post second eye implantation)
Population: This analysis population included all subjects with successful bilateral IOL implantation (Full Analysis Set). Number analyzed is the number of subjects with data available for analysis at specified defocus.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  +2.0 D: number analyzed (Participants) | 43
  +2.0 D | 0.539 (0.1188)
  +1.5 D: number analyzed (Participants) | 43
  +1.5 D | 0.364 (0.1241)
  +1.0 D | 0.213 (0.1339)
  +0.5 D | 0.054 (0.0977)
  0.0 D | -0.049 (0.0697)
  -0.5 D | 0.030 (0.0701)
  -1.0 D | 0.092 (0.0854)
  -1.5 D | 0.060 (0.0917)
  -2.0 D | 0.027 (0.0648)
  -2.5 D | 0.058 (0.0800)
  -3.0 D | 0.134 (0.0850)
  -3.5 D | 0.238 (0.0987)
  -4.0 D | 0.377 (0.1178)
  -4.5 D | 0.510 (0.1367)
  -5.0 D: number analyzed (Participants) | 43
  -5.0 D | 0.604 (0.1222)

2. Secondary Outcome: Binocular Defocus Curve at Month 1
Description: The defocus curve (an indicator of the expected range of vision with a presbyopia-correcting IOL) was tested binocularly (both eyes together) with the subject's best distance correction across full range varied from +2.0 diopter (D) to -5.0 D in 0.5 D increments. VA at each spherical power was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation)
Population: Full Analysis Set. Number analyzed is the number of subjects with data available for analysis at specified defocus.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  +2.0 D: number analyzed (Participants) | 43
  +2.0 D | 0.581 (0.1689)
  +1.5 D: number analyzed (Participants) | 43
  +1.5 D | 0.427 (0.1568)
  +1.0 D: number analyzed (Participants) | 43
  +1.0 D | 0.275 (0.1325)
  +0.5 D: number analyzed (Participants) | 43
  +0.5 D | 0.111 (0.1420)
  0.0 D: number analyzed (Participants) | 43
  0.0 D | -0.015 (0.0815)
  -0.5 D: number analyzed (Participants) | 43
  -0.5 D | 0.049 (0.0785)
  -1.0 D: number analyzed (Participants) | 43
  -1.0 D | 0.086 (0.0678)
  -1.5 D: number analyzed (Participants) | 43
  -1.5 D | 0.093 (0.0800)
  -2.0 D: number analyzed (Participants) | 43
  -2.0 D | 0.080 (0.1046)
  -2.5 D: number analyzed (Participants) | 43
  -2.5 D | 0.090 (0.1229)
  -3.0 D: number analyzed (Participants) | 43
  -3.0 D | 0.167 (0.1253)
  -3.5 D: number analyzed (Participants) | 43
  -3.5 D | 0.264 (0.1455)
  -4.0 D: number analyzed (Participants) | 43
  -4.0 D | 0.360 (0.1385)
  -4.5 D: number analyzed (Participants) | 43
  -4.5 D | 0.505 (0.1585)
  -5.0 D: number analyzed (Participants) | 43
  -5.0 D | 0.640 (0.1358)

3. Secondary Outcome: Binocular Best Corrected Distance Visual Acuity (BCDVA) [4 Meters (m)]
Description: VA was tested binocularly under photopic conditions using the correction obtained from the manual manifest refraction and 100% contrast, ETDRS charts at a distance of 4 meters from the spectacle plane. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set. Number analyzed is the number of subjects with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  Month 1: number analyzed (Participants) | 43
  Month 1 | -0.015 (0.0815)
  Month 3 | -0.049 (0.0697)

4. Secondary Outcome: Monocular Uncorrected Distance Visual Acuity (UCDVA) (4 m)
Description: VA was tested monocularly (each eye separately) under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 4 m from the eye, corresponding to a far distance for visual tasks. UCDVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. Both eyes contributed to the analysis. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: This analysis population included all subjects with successful implantation of the test product in at least one eye (All-implanted Analysis Set). Number analyzed is the number of subjects/eyes with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- TFNT00 First Eye: AcrySof IQ PanOptix Multifocal IOL Model TFNT00 implanted in the capsular bag following cataract removal. Implantation in the first eye
- TFNT00 Second Eye: AcrySof IQ PanOptix Multifocal IOL Model TFNT00 implanted in the capsular bag following cataract removal. Implantation in the second eye
Arm/Group | TFNT00 First Eye | TFNT00 Second Eye
Number analyzed (Participants) | 45 | 44
Number analyzed (Eyes) | 45 | 44
logMAR
  Month 1: number analyzed (Participants) | 43 | 43
  Month 1: number analyzed (Eyes) | 43 | 43
  Month 1 | 0.089 (0.1203) | 0.097 (0.1078)
  Month 3: number analyzed (Participants) | 44 | 44
  Month 3: number analyzed (Eyes) | 44 | 44
  Month 3 | 0.073 (0.1002) | 0.081 (0.1328)

5. Secondary Outcome: Monocular Uncorrected Intermediate Visual Acuity (UCIVA) [60 Centimeters (cm)]
Description: VA was tested monocularly under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 60 cm from the eye, representative of intermediate distances for visual tasks. UCIVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. Both eyes contributed to the analysis. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: All-implanted Analysis Set. Number analyzed is the number of subjects/eyes with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | TFNT00 First Eye | TFNT00 Second Eye
Number analyzed (Participants) | 45 | 44
Number analyzed (Eyes) | 45 | 44
logMAR
  Month 1: number analyzed (Participants) | 44 | 44
  Month 1: number analyzed (Eyes) | 44 | 44
  Month 1 | 0.080 (0.1493) | 0.080 (0.1407)
  Month 3: number analyzed (Participants) | 44 | 44
  Month 3: number analyzed (Eyes) | 44 | 44
  Month 3 | 0.054 (0.1217) | 0.035 (0.1295)

6. Secondary Outcome: Monocular Uncorrected Near Visual Acuity (UCNVA) (40 cm)
Description: VA was tested monocularly under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 40 cm from the eye, representative of near distances for visual tasks. UCNVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. Both eyes contributed to the analysis. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | TFNT00 First Eye | TFNT00 Second Eye
Number analyzed (Participants) | 45 | 44
Number analyzed (Eyes) | 45 | 44
logMAR
  Month 1: number analyzed (Participants) | 44 | 44
  Month 1: number analyzed (Eyes) | 44 | 44
  Month 1 | 0.116 (0.1284) | 0.104 (0.1219)
  Month 3: number analyzed (Participants) | 44 | 44
  Month 3: number analyzed (Eyes) | 44 | 44
  Month 3 | 0.089 (0.1334) | 0.091 (0.1226)

7. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity (UCDVA) (4 m)
Description: VA was tested binocularly under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 4 m from the eye, corresponding to a far distance for visual tasks. UCDVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set. Number analyzed is the number of subjects with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  Month 1: number analyzed (Participants) | 43
  Month 1 | 0.049 (0.1071)
  Month 3 | 0.026 (0.0987)

8. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity (UCIVA) (60 cm)
Description: VA was tested binocularly under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 60 cm from the eye, representative of intermediate distances for visual tasks. UCIVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  Month 1 | 0.015 (0.1242)
  Month 3 | -0.025 (0.1113)

9. Secondary Outcome: Binocular Uncorrected Near Visual Acuity (UCNVA) (40 cm)
Description: VA was tested binocularly under photopic conditions without visual correction using 100% contrast ETDRS charts at a distance of 40 cm from the eye, representative of near distances for visual tasks. UCNVA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 (Day 30-60 post second eye implantation) and Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00
Number analyzed (Participants) | 44
logMAR
  Month 1 | 0.047 (0.1221)
  Month 3 | 0.029 (0.1222)

10. Secondary Outcome: Binocular Photopic Best Corrected Contrast Sensitivity With Glare
Description: Contrast sensitivity (i.e., the ability to detect objects by distinguishing them from their background) was assessed binocularly under photopic conditions at a distance of 8 feet from the eye at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd) using the Vector Vision CSV 1000-HGT with a glare source. A higher numeric value will represent better contrast sensitivity. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log unit
Arm/Group | TFNT00
Number analyzed (Participants) | 44
log unit
  3 cpd | 1.673 (0.1316)
  6 cpd | 1.907 (0.1691)
  12 cpd | 1.539 (0.2113)
  18 cpd | 1.139 (0.2038)

11. Secondary Outcome: Binocular Photopic Best Corrected Contrast Sensitivity Without Glare
Description: Contrast sensitivity (i.e., the ability to detect objects by distinguishing them from their background) was assessed binocularly under photopic conditions at a distance of 8 feet from the eye at spatial frequencies of 3, 6, 12, and 18 cpd using the Vector Vision CSV 1000-HGT without a glare source. A higher numeric value will represent better contrast sensitivity. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log unit
Arm/Group | TFNT00
Number analyzed (Participants) | 44
log unit
  3 cpd | 1.676 (0.1647)
  6 cpd | 1.878 (0.1747)
  12 cpd | 1.588 (0.2317)
  18 cpd | 1.133 (0.2268)

12. Secondary Outcome: Percentage of Subjects Who Responded to Subjective Symptoms Questions (SSQs)
Description: Subjects responded to 12 SSQs based on their experience during past 7 days for quality of vision and any change since cataract surgery as follows; Q1:How satisfied are you with your vision for seeing objects at near distance(ND)? Q2:How often do you wear eyeglasses or contact lenses for seeing objects at ND? Q3:How satisfied are you with your vision for seeing objects at intermediate distance(ID)? Q4:How often do you wear eyeglasses or contact lens for seeing objects at ID? Q5:How satisfied are you with your vision for seeing objects at distance(D)? Q6:How often do you wear eyeglasses or contact lens for seeing objects at D? Q7:How often do you experience halos? Q8:How severe were these halos? Q9:If you CURRENTLY DRIVE: how much difficulty do you have driving at night? Q10:If you DO NOT DRIVE at night, what is the reason? Q11:How satisfied are you with your cataract surgery result? Q12:Would you recommend cataract surgery and new lenses that were put into your eyes to other people?
Time Frame: Preoperative and Month 3 (Day 90-120 post second eye implantation)
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of subjects
Groups:
- TFNT00 Preoperative: All subjects in FAS prior to initiation of treatment
- TFNT00 Month 3: All subjects in FAS who responded at Month 3
Arm/Group | TFNT00 Preoperative | TFNT00 Month 3
Number analyzed (Participants) | 44 | 44
percentage of subjects
  Q1: Very dissatisfied | 47.7 | 2.3
  Q1: Dissatisfied | 40.9 | 4.5
  Q1: Neither satisfied nor dissatisfied | 6.8 | 9.1
  Q1: Satisfied | 4.5 | 63.6
  Q1: Very satisfied | 0.0 | 20.5
  Q2: None of the time | 15.9 | 84.1
  Q2: Some of the time | 15.9 | 13.6
  Q2: Most of the time | 25.0 | 0.0
  Q2: All of the time | 43.2 | 2.3
  Q3: Very dissatisfied | 25.0 | 2.3
  Q3: Dissatisfied | 61.4 | 9.1
  Q3: Neither satisfied nor dissatisfied | 6.8 | 11.4
  Q3: Satisfied | 6.8 | 56.8
  Q3: Very satisfied | 0.0 | 20.5
  Q4: None of the time | 20.5 | 90.9
  Q4: Some of the time | 27.3 | 6.8
  Q4: Most of the time | 25.0 | 0.0
  Q4: All of the time | 27.3 | 2.3
  Q5: Very dissatisfied | 20.5 | 2.3
  Q5: Dissatisfied | 43.2 | 6.8
  Q5: Neither satisfied nor dissatisfied | 25.0 | 20.5
  Q5: Satisfied | 11.4 | 59.1
  Q5: Very satisfied | 0.0 | 11.4
  Q6: None of the time | 31.8 | 95.5
  Q6: Some of the time | 20.5 | 2.3
  Q6: Most of the time | 11.4 | 0.0
  Q6: All of the time | 36.4 | 2.3
  Q7: None of the time | 22.7 | 6.8
  Q7: Some of the time | 45.5 | 25.0
  Q7: Most of the time | 22.7 | 34.1
  Q7: All of the time | 9.1 | 34.1
  Q8: None | 20.5 | 6.8
  Q8: Mild | 29.5 | 11.4
  Q8: Moderate | 34.1 | 50.0
  Q8: Severe | 15.9 | 31.8
  Q9: No difficulty at all | 11.4 | 9.1
  Q9: A little difficulty | 11.4 | 11.4
  Q9: Moderate difficulty | 29.5 | 25.0
  Q9: Extreme difficulty | 25.0 | 22.7
  Q9: NA : I do not drive at night | 22.7 | 31.8
  Q10: Because of your current eyesight | 27.3 | 25.0
  Q10: Because you are not interested in driving | 11.4 | 11.4
  Q10: Because you have other reasons | 22.7 | 27.3
  Q10: NA: I drive at night | 38.6 | 36.4
  Q11: Very dissatisfied | NA — Q11 was not applicable for subjects in Preoperative arm. | 4.5
  Q11: Dissatisfied | NA — Q11 was not applicable for subjects in Preoperative arm. | 2.3
  Q11: Neither satisfied nor dissatisfied | NA — Q11 was not applicable for subjects in Preoperative arm. | 18.2
  Q11: Satisfied | NA — Q11 was not applicable for subjects in Preoperative arm. | 54.5
  Q11: Very satisfied | NA — Q11 was not applicable for subjects in Preoperative arm. | 20.5
  Q12: No | NA — Q12 was not applicable for subjects in Preoperative arm. | 36.4
  Q12: Yes | NA — Q12 was not applicable for subjects in Preoperative arm. | 63.6

ADVERSE EVENTS:
Time Frame: Pre-operation through study completion, an average of 7 months
Description: Adverse Event (AE) was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. Safety Analysis Set. "At Risk" population of preoperative and systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Preoperative: All subjects in the safety analysis set prior to initiation of treatment
- TFNT00 Systemic: All subjects with attempted test article implantation (successful or aborted after contact with the eye)
Arm/Group | Preoperative | TFNT00 First Eye | TFNT00 Second Eye | TFNT00 Systemic
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 1/44 | 2/45
Other Adverse Events (participants affected / at risk) | 1/45 | 23/45 | 20/44 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=45) | TFNT00 First Eye (N=45) | TFNT00 Second Eye (N=44) | TFNT00 Systemic (N=45)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=45) | TFNT00 First Eye (N=45) | TFNT00 Second Eye (N=44) | TFNT00 Systemic (N=45)
Dry eye (Eye disorders) | 0 | 11 | 10 | 0
Glare (Eye disorders) | 0 | 10 | 9 | 0
Visual impairment (Eye disorders) | 1 | 3 | 3 | 0
Halo vision (Eye disorders) | 0 | 3 | 3 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 3 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03268746/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03268746/SAP_001.pdf